CLINICAL TRIAL: NCT01960829
Title: A Single-armed, Open-labeled and Single-centered Phase II Trial of Everolimus in Selected Patients With Metastatic Melanoma: Efficacy and Safety Study
Brief Title: Everolimus in Selected Patients With Metastatic Melanoma: Efficacy and Safety Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Lu Si, Beijing Cancer Hospital Department of Renal Cancer and Melanoma, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001CCN28T
Record Dates: First submitted 2013-09-24; First posted 2013-10-11 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Melanoma; TOR Serine-Threonine Kinases; Neoplasm Metastasis
Keywords: melanoma; TOR Serine-Threonine Kinases
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
This is a single-armed, open-labeled and single-centered study of everolimus in selective patients with metastatic melanoma for evaluation of the efficacy and safety. The study objective is to evaluate efficacy profile of everolimus.

The patients who comply with the inclusion and exclusion criteria will be enrolled. The estimated recruiting duration is 18 months. Everolimus will be given in the dose of 10 mg orally each day at lease 6 months unless disease progression or intolerance. The follow-up is till death(at least 1 year).

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of metastases melanoma. Must have evidence of mutations(Kinase domain) of mTOR . Must be ECOG performance status 0,1, or 2 . Must be estimated life expectancy of 3 months or greater. Must be age 18 years or older, male or female. Must have at least one measurable site of disease as defined by at least 1 cm in greatest dimension.

Adequate organ function. Must be willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

Prior systemic therapy for metastatic disease within 4 weeks. Second malignancy within the last 5 years. Severe and/or uncontrolled medical disease. Received RAD001 or other mTOR inhibitors previously . Hypersensitivity to everolimus Current treatment on another clinical trial. Pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
To assess the progression-free survival (PFS) after treatment with everolimus in selected patients with metastatic melanoma (with mTOR mutation). | 18 months

SECONDARY OUTCOMES:
To assess the overall survival (OS) after treatment with everolimus in selected patients with metastatic melanoma (with mTOR mutation). | 18 months
To evaluate the safety of and tolerability to everolimus in Chinese melanoma patients. | 18 months
To evaluate the quality of life. Strategic goal: Explore and Capitalize on New Indications. | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- LuSi, Beijing, Beijing Municipality, China